CLINICAL TRIAL: NCT04157881
Title: Impact of Rabeprazole-induced Elevated Gastric pH on APO-Dabigatran Exposure in Healthy Volunteers
Brief Title: A Study on the Impact of Rabeprazole-induced Elevated Stomach pH on APO-Dabigatran Exposure in Healthy Volunteers
Acronym: TADA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: TADA_1910_V1.9
Record Dates: First submitted 2019-11-01; First posted 2019-11-08 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2021-03

CONDITIONS: Atrial Fibrillation; Venous Thromboembolism
MeSH Terms: conditions — Atrial Fibrillation; Venous Thromboembolism | interventions — Rabeprazole; Tablets, Enteric-Coated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APO-Dabigatran (Other): Single dose 150mg APO-Dabigatran given with 24 hours of Pharmacokinetic (PK) testing post dose
  Interventions: Drug: APO-Dabigatran 150mg
- APO-Dabigatran and Rabeprazole (Other): 4-7 doses of rabeprazole followed by single dose 150mg APO-Dabigatran given with 24 hours of Pharmacokinetic (PK) testing post dose
  Interventions: Drug: RABEprazole 20 Mg Oral Delayed Release Tablet; Drug: APO-Dabigatran 150mg

INTERVENTIONS:
Drug: RABEprazole 20 Mg Oral Delayed Release Tablet — Absorption of APO-Dabigatran measured with and without influence of rabeprazole
  Arms: APO-Dabigatran and Rabeprazole
Drug: APO-Dabigatran 150mg — Absorption of APO-Dabigatran post single dose

SUMMARY:
Open-label, crossover study recruiting 46 healthy male volunteers comparing the absorption of APO-dabigatran 150 mg per oral (PO) in the absence or presence of a proton pump inhibitor. Participants will serve as their own control when comparing dabigatran exposure in the absence or presence of the proton pump inhibitor, Rabeprazole 20 mg.

DETAILED DESCRIPTION:
Non-valvular atrial fibrillation (AF) and venous thromboembolism (VTE) affect hundreds of thousands of Canadians and many millions worldwide. Affected patients are routinely treated with oral anticoagulants. Vitamin K antagonists (VKAs) were the only orally available anticoagulants for more than 60 years. Over the past decade, Direct Acting Oral Anticoagulants (DOACs) have increasingly replaced VKAs for treatment of patients with AF or VTE because of similar or superior efficacy and safety, and greater convenience. One of these new agents, dabigatran etexilate, has now come off patent in Canada, and at least one generic made by Apotex has been approved by Health Canada.

Prior to their introduction into clinical use, the development of an orally active direct thrombin inhibitors (DTIs) proved technically difficult because it required the conversion of a small, water soluble, poorly absorbable, active site-directed molecule into a fat-soluble prodrug that is transformed back to the active drug after intestinal absorption. In the case of dabigatran, this was achieved by administering it as an oral prodrug, dabigatran etexilate. When administered as the pro-drug, the bioavailability of dabigatran is pH-dependent and is optimal at low pH. To overcome the issue with pH-dependency of drug absorption, dabigatran capsules contain drug pellets, which are made up of a tartaric acid core coated with dabigatran etexilate, thereby maintaining an acid micro-environment (1, 2). After absorption the prodrug is metabolized to the active form dabigatran through esterases that are ubiquitous in the body.

Many patients taking oral anticoagulants are elderly and have an increased gastric pH (3), often as a result of commonly prescribed co-medications such as proton pump inhibitors (PPIs). Optimization of the formulation of originator Pradaxa® (dabigatran etexilate) provides consistent absorption in elderly patients, independent of gastric pH (1, 4), as was demonstrated in phase III trials where consistent outcomes were achieved in the young and elderly, and in the presence and absence of PPI therapy(5).

Generic formulations of dabigatran etexilate are required to demonstrate bioequivalence to the originator in healthy volunteers in order to receive regulatory approval in Canada. According to Canadian regulations and Health Canada, bioequivalence trials do not usually require testing in older patients with an altered gastric pH or in patients taking a PPI (6). The sophisticated pharmaceutical formulation of Pradaxa® ensures stable and reliable absorption despite its low solubility under elevated pH. Pradaxa® has a bioavailability of 6.5% (4, 7) and even any seemingly small alteration in absorption resulting from a change in formulation may significantly affect drug levels. Lower drug levels could lead to an increase in thrombotic events, and higher drug levels could increase bleeding. The European Union (EU) product specific guideline for dabigatran etexilate, however, does require additional bioequivalence studies with elevated gastric pH by means of PPI pre-treatment(8).

APO-Dabigatran is one of the first generic formulations of dabigatran etexilate to be introduced into the Canadian market. APO-Dabigatran compared with Pradaxa® demonstrated similar bioavailability in healthy volunteers, fulfilling the requirements as a generic alternative to the original compound. Unlike Pradaxa®, APO-Dabigatran is formulated using fumaric acid and it is unclear whether this produces a similar pharmacokinetic profile to that of Pradaxa in patients with altered gastric pH, for example in the elderly or those taking a PPI.

This study objective is to determine in healthy volunteers whether concomitant PPI therapy impairs absorption of APO-dabigatran 150 mg and thereby reduces drug blood levels.

ELIGIBILITY:
Inclusion Criteria:

1. 20 to 40 years old
2. Body mass index 18-30 kg/m2
3. Male. Those able to father a child must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information sheet.

Exclusion Criteria:

1. Any documented history of heart, lung, liver, kidney, gastrointestinal, genitourinary, musculoskeletal or endocrine disorders or other systemic illness not specifically listed.
2. Regular use of any medications or herbal supplements/remedies (e.g. St. John's wort).
3. Laboratory values outside of reference range that may compromise safety or validity of the trial.
4. Smoking or alcohol consumption such that the investigators feel that they will not be able to comply with the trial protocol.
5. Measures at screening outside of the reference ranges for systolic and diastolic blood pressure (>140/90) and pulse rate (>90/min).
6. Patients who are not expected to comply with the protocol requirements or not expected to complete the trial as scheduled (includes any condition that, in the investigator's opinion, makes the patient an unreliable trial participant).
7. Previous enrollment in this trial.
8. Currently enrolled in another investigational device or drug trial, or less than 30 days since ending another investigational device or drug trial(s), or receiving other investigational treatment(s)

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
24-hour APO-Dabigatran exposure by peak concentration | 24 Hours
  As measured by peak concentration (Cmax)
24-hour APO-Dabigatran exposure | 24 Hours
  As measured by area under the curve (AUC)

SECONDARY OUTCOMES:
Area under the curve Dilute Thrombin time (dTT) | 24 hours
  dilute thrombin time measured at 0 minutes, 30 minutes, 60 minutes, 90 minutes, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 24 hours to calculate AUC and maximum
Maximum Dilute Thrombin time (dTT) | 24 hours
  dilute thrombin time measured at 0 minutes, 30 minutes, 60 minutes, 90 minutes, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 24 hours to calculate AUC and maximum
Area under the curve activated partial thromboplastin time (aPTT) | 24 hours
  activated partial thromboplastin time measured at 0 minutes, 30 minutes, 60 minutes, 90 minutes, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 24 hours to calculate AUC and maximum
Maximum activated partial thromboplastin time (aPTT) | 24 hours
  activated partial thromboplastin time measured at 0 minutes, 30 minutes, 60 minutes, 90 minutes, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 24 hours to calculate AUC and maximum

CONTACTS AND LOCATIONS:
Overall Officials: John Eikelboom, MBBS, MSc, Principal Investigator — Population Health Research Institute
Locations (1):
- The Population Health Research Institute, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Stangier J. Clinical pharmacokinetics and pharmacodynamics of the oral direct thrombin inhibitor dabigatran etexilate. Clin Pharmacokinet. 2008;47(5):285-95. doi: 10.2165/00003088-200847050-00001. PMID 18399711
- [Background] Coppens M, Eikelboom JW, Gustafsson D, Weitz JI, Hirsh J. Translational success stories: development of direct thrombin inhibitors. Circ Res. 2012 Sep 14;111(7):920-9. doi: 10.1161/CIRCRESAHA.112.264903. PMID 22982873
- [Background] Hurwitz A, Brady DA, Schaal SE, Samloff IM, Dedon J, Ruhl CE. Gastric acidity in older adults. JAMA. 1997 Aug 27;278(8):659-62. PMID 9272898
- [Background] Sarah S. The pharmacology and therapeutic use of dabigatran etexilate. J Clin Pharmacol. 2013 Jan;53(1):1-13. doi: 10.1177/0091270011432169. Epub 2013 Jan 24. PMID 23400738
- [Background] Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, Pogue J, Reilly PA, Themeles E, Varrone J, Wang S, Alings M, Xavier D, Zhu J, Diaz R, Lewis BS, Darius H, Diener HC, Joyner CD, Wallentin L; RE-LY Steering Committee and Investigators. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009 Sep 17;361(12):1139-51. doi: 10.1056/NEJMoa0905561. Epub 2009 Aug 30. PMID 19717844
- [Background] Weitz JI, Earl KM, Leblanc K, Semchuk W, Jamali F. Establishing Therapeutic Equivalence of Complex Pharmaceuticals: The Case of Dabigatran. Can J Cardiol. 2018 Sep;34(9):1116-1119. doi: 10.1016/j.cjca.2018.05.023. Epub 2018 Jun 5. PMID 30093297
- See also: Inc. A. APO-dabigatran Product Monograph. — http://pdf.hres.ca/dpd_pm/00043971.PDF
- See also: Dabigatran etexilate hard capsule 75mg, 110mg, 150mg product-specific bioequivalence guidanc — https://www.ema.europa.eu/en/documents/scientific-guideline/dabigatran-etexilate-hard-capsule-75-mg-110-mg-150-mg-product-specific-bioequivalence-guidance_en.pdf